CLINICAL TRIAL: NCT07380074
Title: The Impact of Physical Activity and Exercise Habits on Mental Health in Medical Residents: Associations With Anxiety, Depression, and Burnout - a Cross-sectional Study
Brief Title: Mental Health Outcomes and Variations in Exercise in Residents
Acronym: MOVE-Res
Status: Completed | Type: Observational
Sponsor: University Hospital, Caen (Other)
Responsible Party: Principal Investigator, Joffrey DRIGNY, Associate Professor, University Hospital, Caen
Other Study IDs: MOVE-Res
Record Dates: First submitted 2026-01-16; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Burnout; Anxiety; Depression Anxiety Disorder; Physical Activity and Wellbeing; Resident Physicians
MeSH Terms: conditions — Burnout, Psychological; Anxiety Disorders; Motor Activity | interventions — Exercise

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- French medical residents
  Interventions: Diagnostic Test: Physical Activity and Mental Health Outcomes Assessment

INTERVENTIONS:
Diagnostic Test: Physical Activity and Mental Health Outcomes Assessment — This observational assessment examines physical activity levels and changes in exercise habits, along with mental health outcomes, in medical residents using validated questionnaires for physical activity, anxiety, depression, and burnout.

SUMMARY:
The goal of this observational study is to learn about the relationship between physical activity levels and mental health outcomes in French medical residents. The main questions it aims to answer are:

Do lower physical activity levels or reductions in exercise since medical school relate to higher anxiety, depression, and burnout among medical residents? Do these associations differ by gender or training-related factors?

Participants will complete online questionnaires assessing their physical activity, changes in exercise habits since medical school, and symptoms of anxiety, depression, and burnout at a single point in time.

ELIGIBILITY:
Inclusion Criteria:

* Medical residents currently enrolled in a French residency program
* Age ≥ 18 years
* Able to provide informed consent
* Willing to complete online questionnaires on physical activity and mental health

Exclusion Criteria:

* Inability to complete questionnaires due to language or cognitive barriers
* Refusal or inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population includes medical residents of all specialties at the University of Caen Normandy in Caen, France. Participants are primarily young adults, both male and female, across different years of residency. They are willing and able to complete online questionnaires assessing physical activity, changes in exercise habits since medical school, and mental health outcomes (anxiety, depression, and burnout).
Sampling Method: Non-Probability Sample
Enrollment: 206 (Actual)
Dates: Start 2022-12-03 (Actual); Primary Completion 2023-05-08 (Actual); Study Completion 2023-09-06 (Actual)

PRIMARY OUTCOMES:
Mental Health Outcomes (Anxiety and Depression) | At study enrollment during residency training (baseline)
  Anxiety and depression in medical residents are assessed using the Hospital Anxiety and Depression Scale (HADS).
  Score Range: 0-21 for each subscale Interpretation: Higher scores indicate greater anxiety or depressive symptoms
Mental Health Outcomes (Burnout) | At study enrollment during residency training (baseline)
  Burnout in medical residents is measured using the Maslach Burnout Inventory (MBI), including emotional exhaustion, depersonalization, and personal accomplishment.
  Emotional Exhaustion: 0-54 (higher scores indicate greater burnout) Depersonalization: 0-30 (higher scores indicate greater burnout) Personal Accomplishment: 0-48 (lower scores indicate greater burnout)
Physical Activity Levels | At study enrollment during residency training (baseline)
  Physical activity in medical residents is assessed using the International Physical Activity Questionnaire (IPAQ), capturing current activity levels and changes in exercise habits since medical school. Levels are categorized as low, moderate, or high and analyzed in relation to mental health outcomes.
  Outcome: Total physical activity expressed in MET-minutes/week Categories: Low, Moderate, High physical activity Interpretation: Higher values indicate greater physical activity
Sport Participation Frequency | At study enrollment during residency training (baseline)
  Participants report the frequency of sport or exercise participation during residency, measured as the number of exercise sessions per week.
Sport Participation Duration | At study enrollment during residency training (baseline)
  Participants report the average duration of exercise sessions during residency. Unit of Measure: Minutes per exercise session
Type of Sport | At study enrollment during residency training (baseline)
  Participants report the type of exercise, both during medical school and residency.
Satisfaction With Current Physical Activity Level (Self-Reported Questionnaire) | At study enrollment during residency training (baseline)
  Satisfaction with current physical activity level is assessed using a self-reported study questionnaire. Participants indicate whether they are satisfied or not satisfied with their current level of physical activity.
  Outcome Measure: Satisfaction with physical activity (Satisfied, Not satisfied)
Change in Physical Activity Level Since Medical School (Self-Reported Questionnaire) | At study enrollment during residency training (baseline)
  Changes in physical activity level since medical school are assessed using a self-reported study questionnaire. Participants indicate whether their current level of physical activity has increased, decreased, or remained unchanged compared with their activity level during medical school.
  Categorical change in physical activity level (Increased / Decreased / No change)

SECONDARY OUTCOMES:
Gender | At study enrollment during residency training (baseline)
  Participants report their gender (male, female, or other) to examine its association with physical activity levels and mental health outcomes.
Age | At study enrollment during residency training (baseline)
  Participants report their age in years to evaluate potential relationships with physical activity and mental health outcomes.
Marital Status and Children | At study enrollment during residency training (baseline)
  Participants report marital status (single, married, in a relationship) and whether they have children, to assess potential influences on exercise habits and mental health outcomes.
Year of Residency | At study enrollment during residency training (baseline)
  Participants indicate their current year of residency training to explore associations with physical activity and mental health outcomes across different stages of residency.
Specialty | At study enrollment during residency training (baseline)
  Participants report their medical specialty to examine whether specialty-related factors are associated with physical activity patterns and mental health outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Caen Normandy, Caen, France

IPD SHARING:
Plan to Share IPD: Undecided